CLINICAL TRIAL: NCT06617078
Title: Benefit of High-flow Nasal Cannula on Persistent Dyspnea in Interstitial Lung Disease: Randomized Multicentric Cross-over Trial
Brief Title: Benefit of High-flow Nasal Cannula on Persistent Dyspnea in Ild
Acronym: HIGHOXFILD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: APHP210079; IDRCB (Other: 2023-A00378-37)
Record Dates: First submitted 2024-01-02; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-01

CONDITIONS: ILD
Keywords: Chronic breathlessness; ILD; high nasal flow canula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Long-Term Oxygen therapy (LTOT) then High Flow Nasal Therapy (HFNT) (Other): 2 weeks of LTOT then 2 weeks of LTOT+HFNT
  Interventions: Procedure: long-term oxygen therapy (LTOT); Procedure: High Flow Nasal Therapy (HFNT)
- High Flow Nasal Therapy (HFNT) then Long-Term Oxygen therapy (LTOT) (Other): 2 weeks of LTOT+HFNT then 2 weeks of LTOT
  Interventions: Procedure: long-term oxygen therapy (LTOT); Procedure: High Flow Nasal Therapy (HFNT)

INTERVENTIONS:
Procedure: long-term oxygen therapy (LTOT) — Usual care with LTOT for 2 weeks
Procedure: High Flow Nasal Therapy (HFNT) — High Flow Nasal delivered by myAirvo3 (4 hours minimum and during th 3-minute chair rise test, 30L/min, 34°C, identical O2 flow rate as LTOT) for 2 weeks

SUMMARY:
The main purpose of this study is to evaluate the effects of high-flow nasal therapy (HFNT) oxygen compared to long-term oxygen therapy (LTOT) on dyspnea and quality of life in intersititial lung disease patients with chronic respiratory failure and persistent breathlessness in whom LTOT has already been initiated.

DETAILED DESCRIPTION:
The study will be a non-blinded, two-arm, crossover (2 periods of 2 weeks each), randomised controlled superiority multicentre trial comparing the effect of HFNT on persistent dyspnoea in intersititial lung disease patients with chronic respiratory failure as compared to LTOT over a two-week period. The oxygen flow rate with HFNT will be the same as for usual care. The HFNT will be used during the night and during the 3-minute chair rise test, it can be used during the day depending on the patient's needs. During the rest of the time, the LTOT will be used as in usual care. Participants will be randomised to receive (1) 2 weeks of LTOT then 2 weeks of LTOT+HFNT or (2) 2 weeks of LTOT+HFNT then 2 weeks of LTOT. The investigators will determine the effect of HFNT on quality of life and dyspnoea. The investigators will also study the effect of HFNT on secondary outcomes listed below. Each assessment will be performed at the end of each 2-week period. Polysomnography will be optional. The study will be conducted in 42 patients with LTOT suffering from persistent breathlessness.

With a total sample of 38 patients and a crossover design, if the real difference on the Saint George's Respiratory Questionnaire (SGRQ) is 6, the standard deviation of the matched difference is 12.5 and the significance threshold is 5%, a two-tailed Student's t test will have a power of 80% to conclude that the difference is significantly different from 0 (Calculated using PASS 14.0.14, Analysis of a cross-over design using difference).These hypotheses are based on the values observed in the article by Nagata et al. (PMID: 29283682), in patients with Chronic Obstructive Pulmonary Diseaes of the same severity, which reported an improvement in the SGRQ-s of -10.8 (95% CI: -15.3; -6.3, i.e. SD of 12.4) with HFNT administered at night for 6 weeks versus LTOT Another study (PMID: 31308647) reported an improvement of -11.9 (CI95% -17.2; -6.6) after an introduction of HFNT. As the minicmal clinical improvement difference for SGRQ is 4, a difference of 6 is considered was both realistic and clinically relevant. A Student's t test allows a conservative approach compared to the use of a linear mixed-effects model retained for the analysis of the primary endpoint.

To take account of reduced precision due to possible loss of follow-up or study withdrawals, the sample was increased by 10%, i.e. 42 patients: 21 in the HFNT+LTOT then LTOT sequence and 21 in the LTOT then HFNT+LTOT sequence.

ELIGIBILITY:
Inclusion Criteria:

* Intertitial lung disease
* Persistant dyspnea (mMRC≥3)
* Long-term oxygen therapy at least for 3 months

Exclusion Criteria:

* Chronic respiratory disease (COPD, lung cancer)
* Pneumothorax,
* Pneumomediastinum,
* Active smoker,
* Patient on non-invasive ventilation or continuous positive airway pressure (CPAP),
* Pregnancy or breastfeeding,
* Unable to read or understand questionnaires,
* No written consent,
* Patients under guardianship,
* No health assurance coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
SGRQ questionnaire : Saint George's Respiratory Questionnaire (symptom component) | 2 weeks
  Symptom component of SGRQ : Scores range from 0 to 100, with higher scores indicating more limitations.

SECONDARY OUTCOMES:
Dyspnea assessement : dyspnoea-12 | 2 weeks
  Dyspnea-12 score range from 0 to 36, with higher score indicating worse breathlessness
Dyspnea assessement : mMRC: Modified Medical Research Council | 2 weeks
  mMRC score : range frome 0 (low) to 4(high) and assesses the intensity of dyspnea
Dyspnea assessement : MDP: Multidimensional dyspnea profile | 2 weeks
  * Immediate affective score range from 0 to 10 with higher score indicating worse breathlessness
  * Sensory score range from 0 to 50 with higher score indicating worse breathlessness
  * Emotional score range from 0 to 50 with higher score indicating worse breathlessness
Quality of life (SGRQ questionnaire) : S.George's Respiratory Questionnaire | 2 weeks
  * Total score range from 0 to 100 with higher score indicating more limitations
  * Activity subscore range from 0 to 100 with higher score indicating more limitations
  * Impact sub-score range from 0 to 100 with higher score indicating more limitations
Quality of life (K-Bild) : The King's Brief Interstitial Lung Disease (KBILD) questionnaire | 2 weeks
  Total score range from 0 to 100 with lower score indicating more limitations
Quality of life questionnaire (SF12): Short Form 12 | 2 weeks
  Total score range from 0 to 100 with higher score indicating more limitations
Anxiety-depression (HADS) : Hospital Anxiety and Depression scale | 2 weeks
  * Anxiety sub-score range from 0 to 21 with higher score indicating more severe anxiety
  * Depression sub-scorerange from 0 to 21 with higher score indicating more severe depression
Distance at 6-minutes walk test | 2 weeks
  Length in meters
Dyspnea (Borg score) at the 6-minutes walk test | 2 weeks
  Score range from 0 to 10 with higher score indicating worst breathlessness
Number of rise at the 3-minutes rise chair test | 2 weeks
  Number of rise
Dyspnea (Borg score) at the 3-minutes rise chair test | 2 weeks
  Score range from 0 to 10 with higher score indicating worst breathlessness
Nocturnal capnography | 2 weeks
  Mean PtcCO2
Respiratory rate | Over 2 weeks
  * Mean day-time respiratory rate measured by a wearable tele-monitoring device (breaths/min)
  * Mean night-time respiratory rate measured by a wearable tele-monitoring device (breaths/min)
Heart rate | Over 2 weeks
  * Mean day-time heart rate measured by a wearable tele-monitoring device (beats/min)
  * Mean night-time heart rate measured by a wearable tele-monitoring device (beats/min)
SpO2 | Over 2 weeks
  * Mean day-time SpO2 measured by a wearable tele-monitoring device (%)
  * Mean night-time SpO2 measured by a wearable tele-monitoring device (%)
Rest | Over 2 weeks
  Mean daily rest hours measured by a wearable tele-monitoring device (hours/day)
Activity | Over 2 weeks
  Mean daily walking hours measured by a wearable tele-monitoring device (hours/day)
Activity | Over 2 weeks
  Mean daily steps measured by a wearable tele-monitoring device (steps/day)
Sleep Quality only in patients for whom nocturnal polysomnography is performed during one night (optional) | 2 weeks
  Sleep duration (minutes)
Sleep Quality only in patients for whom nocturnal polysomnography is performed during one night (optional) | 2 weeks
  Onset latency (minutes)
Sleep Quality only in patients for whom nocturnal polysomnography is performed during one night (optional) | 2 weeks
  Percentage of REM sleep (%)
Sleep Quality only in patients for whom nocturnal polysomnography is performed during one night (optional) | 2 weeks
  Sleep efficiency (%)
Sleep Quality only in patients for whom nocturnal polysomnography is performed during one night (optional) | 2 weeks
  Apnoea-hypopnoea index (per hour)
Sleep Quality only in patients for whom nocturnal polysomnography is performed during one night (optional) | 2 weeks
  Index of arousal and micro-arousals (per hour)
Sleep Quality only in patients for whom nocturnal polysomnography is performed during one night (optional) | 2 weeks
  Time spent at SpO2 below 90% (TST90) (%)
Acute exacerbation and/or increase in resting oxygen flow | 2 weeks
  Number of patients with (i) an acute exacerbation defined as the onset or acute worsening of dyspnoea, associated with an increase in radiological lesions (new ground-glass opacities and/or bilateral condensations) not explained by heart failure or overload, or (ii) an increase in resting oxygen flow of more than 2 L/min (on medical prescription).
HFNT(High Flow Nasal Therapy) compliance | 2 weeks
  * Average daily hours of use of the HFNT device
  * Average daily hours of use of LTOT
HFNT (High Flow Nasal Therapy) acceptability | 2 weeks
  Side effects

CONTACTS AND LOCATIONS:
Overall Officials: Capucine Morélot-Panzini, MD,PhD, Prof, Principal Investigator — APHP • Assistance Publique des hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatiqueet des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients. Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.